CLINICAL TRIAL: NCT06928610
Title: A Randomized Controlled Trial of the HeartMath Resilience Program: Exploring the Impact of Stress on Jail Staff Performance and Retention
Brief Title: Heart Math Resilience Program on Jail Staff
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: Leon County Sheriff's Office (Unknown)
Responsible Party: Principal Investigator, Tanya Renn, Principal Investigator, Florida State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00004706; 15PNIJ-23-GG-02231-NIJB (Other Grant/Funding Number: National Institute of Justice (NIJ))
Record Dates: First submitted 2025-04-08; First posted 2025-04-15 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Stress
Keywords: Chronic Stress; Perceptions of job satisfaction; Workplace safety; Occupational stress; Retention and absenteeism; Punitive attitudes; Apprehension to employ use of force; HeartMath; Resiliency-based intervention; Correctional officers
MeSH Terms: conditions — Occupational Stress

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with an intervention arm and a waitlist control arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HeartMath Resilience Program (Experimental): Participants will receive programming alongside their regularly scheduled defensive tactics training.
  Interventions: Behavioral: HeartMath Resilience Program
- Waitlist Control, No Intervention (No Intervention): Participants in the waitlist control group will receive their regularly scheduled training programs

INTERVENTIONS:
Behavioral: HeartMath Resilience Program — Resiliency-based intervention designed to reduce stress, build resilience, and maintain energy levels.
  Other Names: HeartMath
  Arms: HeartMath Resilience Program

SUMMARY:
The study is a multiple cohort, staggered-entry, waitlist randomized controlled trial evaluating the effectiveness of a comprehensive resiliency-based program in reducing stress for correctional officers employed by the Leon County Sheriff's Office in Tallahassee, FL.

DETAILED DESCRIPTION:
The primary objective of the study is to implement and evaluate the effectiveness of a comprehensive resiliency-based intervention, HeartMath, designed to reduce stress for correctional officers (COs) currently employed with the Leon County Sherriff's Office in Tallahassee, Florida. The study will also examine whether the intervention 1) improves perceptions of job satisfaction, workplace safety, and occupational stress; 2) improves CO retention and decreases absenteeism; 3) results in less punitive attitudes and greater apprehension to employ use of force.

ELIGIBILITY:
Inclusion Criteria:

* Leon County Sheriff's Office jail correctional officers.
* Attending a defensive tactics training by Leon County Sheriff's Office
* Age 18 years or older
* Conversational English
* Being willing and cognitively able to provide consent.

Exclusion Criteria:

* Not meeting Inclusion Criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Change In Perceived Chronic Stress Level | Baseline, 3 months, 6 months, 9 months, 12 months
  Utilizing Wheaton Chronic Stress Inventory participants will rate their perceived stress on a three-point Likert scale (0 = "not true," 1 = "somewhat true," and 2 = "very true"). Scores are summed where higher values indicate more exposure to chronic stress. Scores range from 0 to 102.
Change in Perceived Work Stress Level | Baseline, 3 months, 6 months, 9 months, 12 months
  Utilizing the Work Stress scale participants will rate their perceived work stress on a 4-point Likert scale and summed where higher values indicate more exposure to work stress. Response categories range between 1 (strongly disagree) and 4 (strongly agree). Scores range between 14 and 56.

SECONDARY OUTCOMES:
Change in Workplace Safety Perceptions | Baseline, 3 months, 6 months, 9 months, 12 months
  Utilizing a five-item index tapping overall perceptions of the danger of the officer's workplace (e.g., My job is more dangerous than other jobs). Responses are assessed using four response categories ranging from 1 (strongly disagree) to 4 (strongly agree). Scores summed with lower values representing increased perception of safety.
Change in Job Satisfaction | Baseline, 3 months, 6 months, 9 months, 12 months
  Utilizing a five-item scale based on the general scale developed by Brayfield and Rothe and subsequently modified for use with COs. Response categories range from 1 (strongly disagree) to 4 (strongly agree). Scores summed with higher values representing increased levels of job satisfaction.
Change in Support for Punishment | Baseline, 3 months, 6 months, 9 months, 12 months
  Utilizing the Support for Punishment index originally developed by Cullen et al. It is a nine-item self-report index to assess officer attitudes toward punishment and has been used previously to assess CO support for more punitive treatment of incarcerated individuals. Response categories range from 1 (strongly disagree) to 4 (strongly agree). Scores summed with higher values representing greater support for punishment. Scores range from 9 to 36.
Change in Support for Treatment | Baseline, 3 months, 6 months, 9 months, 12 months
  Utilizing the Support for Treatment index developed by Cullen et al. to be used with COs and consists of eight items tapping officer support for a more treatment-oriented approach to corrections. Response categories range from 1 (strongly disagree) to 4 (strongly agree). Higher values representing greater support for treatment. Scores range from 8 to 32.
Change in Readiness to Use Force | Baseline, 3 months, 6 months, 9 months, 12 months
  Utilizing a six-item measure originally developed by Griffin and used previously to assess CO attitudes toward the use of force in commonly encountered situations to assess officers' propensity to use force. Responses are assessed using four response categories ranging from 1 (strongly disagree) to 4 (strongly agree). Higher values representing increased levels of readiness to use force.
Change in Officer Absenteeism | Baseline, 3 months, 6 months, 9 months, 12 months
  Utilizing human resources data provided by LCSO, absenteeism will be measured as the number of days officers called in sick or did not report for a scheduled shift during the study period.
Officer Employment Status | Baseline, 3 months, 6 months, 9 months, 12 months
  Utilizing human resources data provided by LCSO to determine whether an officer was still employed at the end of the study period.
Change in Organizational Committment | Baseline, 3 months, 6 months, 9 months, 12 months
  Utilizing a five-item index tapping officers' connection to their current organization and whether they plan to stay with the organization in the future. Response categories range from 1 (strongly disagree) to 4 (strongly agree). Scores summed with higher values representing increased levels of organizational commitment. Scores range from 5 to 20.
Change in Turnover Intent | Baseline, 3 months, 6 months, 9 months, 12 months
  Utilizing a four-item index originally developed by Lambert and colleagues to assess COs' intentions to leave their current place of employment. Response categories range from 1 (strongly disagree) to 4 (strongly agree). Higher values represent greater intent to change employment. Scores range from 4 to 16.
Change in Views on Absenteeism | Baseline, 3 months, 6 months, 9 months, 12 months
  Utilizing a two-item index adapted from previous measures tapping sick leave use and adapted for use with COs to assess officers' perceptions of missing work. Response categories range from 1 (strongly disagree) to 4 (strongly agree). Higher scores indicate greater willingness to miss work with scores ranging from 2 to 8.

OTHER OUTCOMES:
Change in PTSD | Baseline, 3 months, 6 months, 9 months, 12 months
  Utilizing the 20-item PTSD Checklist for DSM-5 (PCL-5) to assess PTSD symptoms. All items are scored on a five-point Likert scale with 0= "not at all" and 4= "extremely." Scores above 33 indicate current incidence of PTSD.
Change in Depression | Baseline, 3 months, 6 months, 9 months, 12 months
  Utilizing the 11-item major depressive disorder subscale of the MINI International Neuropsychiatric Interview (MINI) to assess current incidence of depression. Items are rated on a dichotomous Yes/No scale and follow DSM-5 psychiatric guidelines.
Change in Anxiety | Baseline, 3 months, 6 months, 9 months, 12 months
  Utilizing the 7-item anxiety subscale of the MINI International Neuropsychiatric Interview (MINI) to assess current anxiety disorders. Items are rated on a dichotomous Yes/No scale and follow psychiatric guidelines of the DSM-5.
Change in Incidence of Substance Use Disorder | Baseline, 3 months, 6 months, 9 months, 12 months
  Utilizing the 9-item substance use disorder subscale of the MINI International Neuropsychiatric Interview (MINI) to assess current incidence of substance use disorders. Items are rated on a dichotomous Yes/No scale and follow psychiatric guidelines of the DSM-5.
Change in Impulsivity | Baseline, 3 months, 6 months, 9 months, 12 months
  Utilizing the Barratt Impulsivity Scale (BIS) to assess general impulsiveness on six first-order factors (attention, motor, self-control, cognitive complexity, perseverance, and cognitive instability impulsiveness) and three second-order factors (attentional, motor, and non-planning impulsiveness). The BIS is composed of 30 items describing common impulsive or non-impulsive (for reverse scored items) behaviors and preferences. Participants select a number on the following scale: 1 if you rarely or never act or think that way, 2 if you occasionally think that way, 3 if you often think that way, or 4 if you almost or always think that way. Scores range from 30 to 120. A higher score indicates greater impulsivity.
Change in Aggression | Baseline, 3 months, 6 months, 9 months, 12 months
  Utilizing the 12-item Brief Aggression Questionnaire (BAQ) to evaluate physical aggression, verbal aggression, anger, and hostility. Scores range from 12 to 60. A higher score indicates greater aggression.
Change in Psychological Distress | Baseline, 3 months, 6 months, 9 months, 12 months
  Utilizing the Brief Symptom Inventory (BSI) to assess symptoms of distress in adults. The BSI is a 53-item self-report screening tool that asks respondents to rate their level of psychological distress over the past seven days based on a five-point Likert scale (0 = "not at all" to 5 = "extremely"). The BSI provides subscale scores on dimensions of somatization, depression, and anxiety as well as a Global Severity Index (GSI) that is calculated based on a sum of all items. Subscale scores range from 0 to 4. Higher scores on the BSI indicate higher levels of symptomology.
Change in Psychological Wellbeing | Baseline, 3 months, 6 months, 9 months, 12 months
  Utilizing the Ryff Psychological Wellbeing Index to assess officer wellbeing. The Ryff is an 18-item self-report tool that asks respondents to indicate how strongly they agree or disagree with 18 statements. Responses are based on a seven-point Likert scale (1 = "strongly agree" to 7 = "strongly disagree"). The Ryff provides subscale scores on dimensions of autonomy, environmental mastery, personal growth, positive relations with others, purpose in life, and self-acceptance as well as a global wellbeing index that is calculated based on a sum of all items. Subscale scores range from 3 to 21 and the global wellbeing scores range from 18 to 126. Higher scores indicate higher levels of wellbeing.

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Renn, PhD, Principal Investigator — Florida State University
Locations (1):
- Leon County Detention Facilities, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) from this clinical trial will be shared in a de-identified format, including demographics, clinical characteristics, and outcomes, in accordance with applicable regulations and ethical guidelines. Data will be made available upon reasonable request after the completion of the trial and publication of primary results, for a period of three years. Access will be granted to qualified researchers affiliated with academic institutions, justice-involved entities, or regulatory bodies. Researchers interested in accessing the data must submit a formal request to trenn@fsu.edu. Upon approval, data will be shared through a secure data repository or other appropriate methods to ensure participant confidentiality. In addition to the IPD, supporting documents such as the study protocol, statistical analysis plan, and informed consent form may also be available upon request.